CLINICAL TRIAL: NCT05163847
Title: Phase 1b Study to Investigate the Safety and Immunogenicity of Cam2020 (A/Cambodia/e0826360/2020) M2SR H3N2 Monovalent Influenza Vaccine Administered Alone or With Licensed, Inactivated Influenza Vaccine in Adults 65 to 85 Years Old
Brief Title: Safety and Immunogenicity of Cam2020 M2SR H3N2 Monovalent Influenza Vaccine Alone or With Licensed IIV in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FluGen Inc (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FLUGEN-H3N2-V006; CDMRP-PR203559 (Other Grant/Funding Number: USAMRAA)
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Subjects assigned randomly to one of four cohorts concurrently
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Syringes wrapped to obscure color of contents
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- M2SR only dose (Experimental): Intranasal M2SR vaccine and intramuscular placebo dose
  Interventions: Biological: Cam2020 M2SR H3N2 influenza vaccine; Other: IM Placebo
- M2SR with IIV dose (Experimental): Intranasal M2SR vaccine and intramuscular IIV dose
  Interventions: Biological: Cam2020 M2SR H3N2 influenza vaccine; Biological: Fluzone HD IIV
- IIV only dose (Active Comparator): Intranasal placebo dose and intramuscular IIV dose
  Interventions: Biological: Fluzone HD IIV; Other: IN Placebo
- Placebo only dose (Placebo Comparator): Intranasal placebo dose and intramuscular placebo dose
  Interventions: Other: IN Placebo; Other: IM Placebo

INTERVENTIONS:
Biological: Cam2020 M2SR H3N2 influenza vaccine — Administered intranasally on Day 1
  Arms: M2SR only dose; M2SR with IIV dose
Biological: Fluzone HD IIV — Administered intramuscularly on Day 1
  Arms: IIV only dose; M2SR with IIV dose
Other: IN Placebo — Administered intranasally on Day 1
  Arms: IIV only dose; Placebo only dose
Other: IM Placebo — Administered intramuscularly on Day 1
  Arms: M2SR only dose; Placebo only dose

SUMMARY:
This is a randomized, double-blind, double-dummy, placebo-controlled Phase 1b study evaluating the safety and immunogenicity of the investigational Cam2020 M2SR H3N2 influenza vaccine delivered IN alone or concomitantly with inactivated influenza vaccine (IIV) delivered IM to a healthy adult population age 65 to 85 years at time of enrollment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, placebo-controlled Phase 1b study evaluating the safety and immunogenicity of the investigational Cam2020 M2SR H3N2 influenza vaccine delivered IN alone or concomitantly with IIV delivered IM to a healthy adult population age 65 to 85 years at time of enrollment. Eligible subjects will be randomized concurrently in a 3:3:3:1 ratio to receive one administration of Cam2020 M2SR alone (Cohort 1, n=90), Cam2020 M2SR along with IIV (Cohort 2, n=90), IIV alone (Cohort 3, n=90), or placebo (Cohort 4, n=30).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to provide written informed consent to participate; a legally authorized representative (LAR) may not be used.
2. Males and nonchildbearing potential females 65-85 years of age at the time of consent.
3. Subjects must be willing to adhere to the requirements of the study and willing and able to communicate with the Investigator and understand the requirements of the study.
4. Healthy adults and those with stable chronic conditions as determined by medical history, physical examination, vital signs, clinical safety laboratory examinations and clinical judgment of the Investigator to be eligible for study inclusion.

Exclusion Criteria:

1. Any acute or chronic physical or mental health condition that would limit the subject's ability to complete the study, increase risk of study participation or participant, or may interfere with interpretation of study results as based on the assessment by the Investigator.
2. Abnormal screening hematology or chemistry value per the US FDA Guidance: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials
3. Currently receiving, or planned to receive during the study, any immunosuppressive therapy.
4. Had a flu-like illness, influenza treatment, or prophylactic influenza viral drug administered in the previous 6 months before investigational product administration.
5. History of receipt of any live virus vaccine within 56 days of study entry, licensed or investigational vaccine within 28 days of Visit 01 or investigational drug within the past 6 months. An exception is made for receipt of a Covid-19 vaccine whether licensed or under EUA as long as the final dose was given at least 28 days prior to Visit 01.
6. Planned receipt of licensed vaccine, other than the study-provided licensed influenza vaccine, during the 28 days following Visit 01 or another investigational vaccine or investigational drug during the study period.
7. Receipt of blood/plasma products or immunoglobulin within 6 months before administration of the investigational product or planned for during the period of study participation.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 303 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Solicited AEs during 7 days after experimental treatment | Day 1 to Day 8
  The number and percentage of subjects who experience solicited local and systemic reactions during the 7 days after vaccine administration of M2SR administration alone or with IIV
Unsolicited AEs during 28 days after experimental treatment | Day 1 to Day 29
  The number and percentage of subjects who experience unsolicited AEs during the 28 days after vaccine administration of M2SR alone or with IIV.
SAEs through 28 days after experimental treatment | Day 1 to Day 29
  The number and percentage of subjects who experience SAEs from the time of informed consent through 28 days after vaccine administration of M2SR alone or with IIV.

CONTACTS AND LOCATIONS:
Overall Officials: Pamuk Bilsel, Study Director — FluGen Inc
Locations (6):
- United States (6):
  - United Medical Research, Port Orange, Florida
  - Velocity Clinical Research, Meridian, Idaho
  - Johnson County Clin Trials, Lenexa, Kansas
  - Rochester Clinical Research, Rochester, New York
  - Velocity Clinical Research, Beechwood, Ohio
  - Velocity Clinical Research, Cedar Park, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eiden J, Fierro C, White A, Davis M, Rhee M, Turner M, Murray B, Herber R, Aitchison R, Marshall D, Moser MJ, Belshe R, Greenberg H, Coelingh K, Kawaoka Y, Neumann G, Bilsel P. Safety and immunogenicity of the intranasal H3N2 M2-deficient single-replication influenza vaccine alone or coadministered with an inactivated influenza vaccine (Fluzone High-Dose Quadrivalent) in adults aged 65-85 years in the USA: a multicentre, randomised, double-blind, double-dummy, phase 1b trial. Lancet Infect Dis. 2024 Oct;24(10):1118-1129. doi: 10.1016/S1473-3099(24)00351-7. Epub 2024 Jul 11. PMID 39004096